CLINICAL TRIAL: NCT00848874
Title: Phase II Study of a Portable Visual Guidance System for Use by AS/HFA Students in Inclusion Settings
Brief Title: Portable Visual Guidance System Phase II
Acronym: PVGS-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minna Levine, PhD (Industry)
Collaborators: SymTrend Inc. (Industry); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor-Investigator, Minna Levine, PhD, Co-Invesetigator, SymTrend Inc.
Organization: SymTrend Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2R41MH075162 (NIH); NIHM_2R41MH75162--02A1
Record Dates: First submitted 2008-04-25; First posted 2009-02-20 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Asperger Syndrome; High Functioning Autism
MeSH Terms: conditions — Asperger Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PVGS User (Experimental)
  Interventions: Behavioral: PVGS

INTERVENTIONS:
Behavioral: PVGS — Student use of SymTrend PVGS daily then tapering off for 14 weeks in conjunction to ratings by a coach.

SUMMARY:
Abstract: In Phase I, we designed and tested a Portable Visual Guidance System (PVGS), which combines a PDA - for user guidance - and an Internet website - for linking the user to an educational support team. Use of the PVGS 1) significantly improved the in vivo social pragmatics of students diagnosed with Aspergers Syndrome/Higher Functioning Autism (AS/HFA); 2) revealed additional ways of improving social pragmatics; and 3) improved activity management in scheduling and vocational tasks.

In Phase II, we will focus on social pragmatics and two closely related skills: feelings management and assignment management. We aim to:

1. Replicate Phase I success in the most educational setting for AS/HFA high school aged students: mainstream school inclusion classes.
2. Replicate Phase I findings more efficiently, with a less highly trained, on-site coaching staff and with more distant (non-site) expert supervision of that staff.
3. Contrast the outcomes of the curriculum with a diagnosis-matched wait-list control group.
4. Develop and implement software that will enable on-site staff to create and modify individualized guidance and monitoring screens as needs arise.
5. Design a commercially attractive package of software, video training, video-conferenced support, and manuals.
6. Complete the translation of the SymTrend website and all the above tools into Spanish.

Significance: Successful completion of Phase II will:

1. Provide a very effective and comprehensive system for teaching social pragmatics and related management skills to AS/HFA persons in an inclusion context.
2. Provide a means of evaluating IEP effectiveness, thereby enabling a better use of special education funds and a reduction of litigation over IEP plan appropriateness and utility.
3. Provide substantial support for our theoretical rationale for curriculum building in Special Education - a rationale that can guide the formulation of IEPs.
4. Provide a theoretical rationale, an intervention framework, and intervention support technology that can be extended to cognitive behavioral treatment of other neuropsychiatric disorders and can be adapted for other forms of healthcare guidance.
5. Provide an investigative system, as well as an intervention system, for tracking behavioral change in studies of frontal lobe and limbic neuroplasticity in neuropsychiatric disorders.

ELIGIBILITY:
Inclusion Criteria:

* Ages 11-21
* Diagnosis of AS/HFA
* A student at participating high school and middle schools (Newton, MA; Brockton, MA; Veritas Christian Academy, Fletcher, NC; Durham, NC.

Exclusion Criteria:

* Participating in another study

Ages: 11 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2008-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Students who use the PVGS will demonstrate improved classroom social pragmatics and executive functioning. | Completion of intervention and three months hence

CONTACTS AND LOCATIONS:
Overall Officials: Gary Mesibov, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Minna Levine, PhD, Study Director — SymTrend Inc.
Locations (1):
- SymTrend, Inc., Belmont, Massachusetts, United States